CLINICAL TRIAL: NCT00918281
Title: A Test-retest Study to Assess Reproducibility of 18F Uptake by Solid Tumors Using PET Imaging Following Intravenous Administration of AH111585 (18F) Injection.
Brief Title: Reproducibility of 18F Uptake by Solid Tumors Using PET Imaging Following Intravenous Administration of (18F) Injection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: BIAFFIN GmbH & Co. KG (Biomolecular Interaction Analyses) (Unknown); Quintiles, Inc. (Industry); i3 Statprobe (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-135-004
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Solid Tumors; High Grade Gliomas; Lung Cancer; Head and Neck Cancer; Sarcoma; Renal Cell Carcinoma; Breast Cancer
MeSH Terms: conditions — Lung Neoplasms; Head and Neck Neoplasms; Sarcoma; Carcinoma, Renal Cell; Breast Neoplasms | interventions — AH 111585; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fluciclatide Injection (Experimental): Fluciclatide Injection
  Interventions: Drug: Fluciclatide Injection

INTERVENTIONS:
Drug: Fluciclatide Injection — Fluciclatide Injection (AH111585 (18F) Injection)
  Other Names: Fluciclatide; AH111585 (18F) Injection

SUMMARY:
Study aimed to assess the reproducibility of PET imaging using AH111585 (18F) Injection. Subjects are evaluable if they undergo 2 administrations of AH111585 (18F) Injection (3 to 8 days apart) and the corresponding PET acquisitions, and tumors demonstrate detectable levels of 18F uptake on PET.

ELIGIBILITY:
Inclusion Criteria:

* The subject has been diagnosed with at least one solid primary or metastatic tumor greater than 2.0 cm in diameter, including but not limited to NSCLC, RCC, GBM, melanoma, sarcoma, breast and H&N cancers.
* The subject has received clinical routine imaging diagnostic work-up within 8 weeks prior to the first [18F]AH111585 PET scan.
* The subject has a clinically acceptable (as judged by the investigator) physical examination at screening and is capable of self-care.

Exclusion Criteria:

* The subject has known hyper- or hypo-coagulation syndromes.
* The subject has received chemotherapy within 3 weeks, or received radiotherapy, surgery or any other treatment against cancer within 4 weeks prior to the first [18F]AH111585 PET scan.
* The subject is scheduled to undergo chemotherapy, radiotherapy, surgery or any other treatment against cancer between the first and second [18F]AH111585 PET scans.
* The subject is scheduled to undergo biopsy for the target tumour between the first and second [18F]AH111585 PET scans.
* The subject has intra-hepatic tumour(s) only.
* For the immuno-histochemistry group, the subject's target tumour has been biopsied less than or equal to 1 week prior to the first [18F]AH111585 PET scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Winick, Ph.D., Principal Investigator — GE Healthcare
Locations (1):
- 101 Carnegie Center, Princeton, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 70 Subjects started and enrolled in this study. 41 Subjects completed this study and 29 did not complete this study.
Pre-assignment Details: Due to the number of subjects that did not complete this study, additional subjects were enrolled bring to total enrolment to 70 subjects.
Groups:
- 1 Fluciclatide Injection: AH111585 (18F) Injection : AH111585 (18F) Injection
Period: Overall Study
Arm/Group | 1 Fluciclatide Injection
Started | 70
Completed | 41
Not Completed | 29
Not completed — Physician Decision | 29

BASELINE CHARACTERISTICS:
Population: 70 Subjects enrolled. A total of 49 subjects received a least one dose of Fluciclatide administration.
Groups:
- 1 Fluciclatide Injection: Fluciclatide Injection (AH111585 (18F) Injection)
Arm/Group | 1 Fluciclatide Injection
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 20
Region of Enrollment [Number; unit: participants]
  India | 18
  Korea, Republic of | 8
  Sweden | 4
  United Kingdom | 19

OUTCOME MEASURES:

1. Primary Outcome: Test Image and Retest Image Reproducibility of Fluciclatide Injection ([18F]AH111585) Uptake by Solid Tumors Following Intravenous Administration of AH111585 (18F) Injection Via PET Imaging.
Description: Mean relative differences of Standardized uptake value (SUV) following intravenous administration of AH111585 (F18) Injection between the two PET imaging sessions.
Time Frame: Forty minutes, 65 minutes and 90 minutes post Fluciclatide administration.
Population: Subjects received 2 doses of Fluciclatide Injection (AH111585 (18F) Injection).
Measure: Mean (Standard Deviation); unit: Standardized Uptake Value
Groups:
- Imaging Session 1: Fluciclatide Injection (AH111585 (18F) Injection) at 10mCi [370 megabecquerels (MBq)]
- Imaging Session 2: Fluciclatide Injection (AH111585 (18F) Injection)
- Relative Difference: The Relative difference between imaging sessions 1 and 2.
Arm/Group | Imaging Session 1 | Imaging Session 2 | Relative Difference
Number analyzed (Participants) | 39 | 39 | 39
Standardized Uptake Value
  40 Minute Post Injection | 4.536 (2.2113) | 4.671 (2.4485) | 0.0198 (0.16099)
  65 Minute Post Injection | 4.584 (2.3266) | 4.675 (2.4489) | 0.0216 (0.17466)
  90 Minute Post Injection | 4.404 (2.2761) | 4.691 (2.6445) | 0.0506 (0.22251)

2. Secondary Outcome: The Safety of Greater Than or Equal to 2 Administrations, Each of a Maximum of 370MBq, Fluciclatide Injection (AH111585 (18F) Injection) in Subjects With Solid Primary or Metastatic Tumors.
Description: Safety was monitored throughout the duration of the subject's participation.
Time Frame: Up to 8 weeks post contrast administration.
Population: The variable is looking at the Overall Summary of Treatment-Emergent Adverse Events (TEAE). Subjects could have experienced more than one TEAE. The category titles refer to Severe Adverse Events(SAE) and Adverse Events (AE).
Measure: Number; unit: number of adverse events
Groups:
- Number of Adverse Events: The number of adverse events in relationship to the categories descrbed using Fluciclatide Injection (AH111585 (18F) Injection).
Arm/Group | Number of Adverse Events
Number analyzed (Participants) | 49
number of adverse events
  Any TEAE | 18
  Total number of TEAEs | 47
  Any TEAE at least related to Drug | 1
  Intesity-Mild | 3
  Intensity-Moderate | 8
  Intensity-Severe | 7
  Any SAEs | 7
  Any SAE at least related to Drug | 0
  Any AE leading to Study Discontinuation | 1
  Any AE leading to Death | 2
  Any AE leading to death at least related to Drug | 0

ADVERSE EVENTS:
Time Frame: Data was collected up to 8 weeks post contrast drug administration.
Arm/Group | 1 Fluciclatide Injection
Serious Adverse Events (participants affected / at risk) | 7/49
Other Adverse Events (participants affected / at risk) | 3/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Fluciclatide Injection (N=49)
Lower respiratory Tract Infection (Infections and infestations) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Carcinoma / Metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Spinal Cord Compression (Nervous system disorders) | 1 (1)
Lymphadenectomy (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Fluciclatide Injection (N=49)
Asthenia (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No